CLINICAL TRIAL: NCT03964558
Title: An Open Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Acebilustat (CTX-4430) in Healthy Male Subjects
Brief Title: Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Acebilustat (CTX-4430)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTX-4430-ADME-101
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Heathy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 100 mg [14C]-acebilustat (Other): a single oral dose of 100 mg [14C]-acebilustat
  Interventions: Drug: [14C]-acebilustat solution

INTERVENTIONS:
Drug: [14C]-acebilustat solution — Acebilustat is a novel synthetic small molecule leukotriene A4 hydrolase (LTA4H) inhibitor.

SUMMARY:
This is a single-centre, open-label, non-randomised, single oral dose study in healthy male subjects. It is planned to enroll and dose 6 subjects. Subjects will be admitted to the clinical unit on the evening of Day 1 prior to investigational medicinal product (IMP) administration. Subjects will be dosed on the morning of Day 1 and it is planned that they will remain resident in the clinic until up to 168 hour after dosing (up to Day 8). It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% or if <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 hour periods.

ELIGIBILITY:
Inclusion Criteria:

• Body mass index of 18.0 to 35.0 kg/m2

Exclusion Criteria:

* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta: amount excreted (Ae) and Ae as a percentage of the administered dose (%Ae), cumulative recovery (CumAe), and cumulative recovery expressed as a percentage of the administered dose (Cum%Ae) | Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No